CLINICAL TRIAL: NCT03812627
Title: Study of Systemic Impact of Trace Elements Release by Implantable Medical Devices. Identification of Biomarkers of Systemic Inflammation
Acronym: PROMETOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP180539
Record Dates: First submitted 2019-01-11; First posted 2019-01-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Biomarker; Systemic Inflammation
Keywords: Implantable medical devices; Biomarker; Systemic inflammation
MeSH Terms: interventions — Blood Specimen Collection; Urination; Autopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Re-intervention of hip prosthesis made of ceramic or metal (Experimental): Re-intervention surgery: blood, urine, hair, synovial fluid and peri-prosthetic tissue collections.
  50 patients for re-intervention of hip prosthesis with friction couples of: ceramic-on-ceramic or metal-on-metal
  (25 patients by group)
  Interventions: Other: Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections
- Re-intervention of hip prosthesis of stainless steel ball (Experimental): Re-intervention surgery: blood, urine, hair, synovial fluid and peri-prosthetic tissue collections.
  50 patients for re-intervention of hip prosthesis of stainless steel ball.
  Interventions: Other: Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections
- Re-intervention of knee prosthesis (Experimental): Re-intervention surgery: blood, urine, hair, synovial fluid and peri-prosthetic tissue collections.
  50 inpatient subjects for re-intervention of knee prosthesis polyethylene-on-metal.
  Interventions: Other: Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections
- Dead patients IMD holders autopsied (Experimental): Autopsy: 80 dead patients IMD holders will be autopsied.
  Interventions: Other: Autopsy
- Dead patients non-IMD holders autopsied (Active Comparator): Autopsy: dead patients non-IMD holders autopsied, 30 subjects in this arm.
  Interventions: Other: Autopsy
- patients before first prosthesis surgery (Active Comparator): Before the initial prosthesis surgery: 30 patients Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections will be done
  Interventions: Other: Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections

INTERVENTIONS:
Other: Blood, urine, hair, synovial fluid and peri-prosthetic tissue collections — All inpatient subjects: following samples will be collected during hospitalization:
  Twice blood and urine collections:
  1. at the beginning of hospitalization: 10 ml of blood + 5 ml of urine;
  2. at the end of hospitalization: 5 ml of blood + 5 ml of urine. Synovial fluid collection: 1 ml Peri-prosthetic tissue collection: about 1 cm3 Hair collection: a single hair of 0.5 cm diameter
  Arms: Re-intervention of hip prosthesis made of ceramic or metal; Re-intervention of hip prosthesis of stainless steel ball; Re-intervention of knee prosthesis; patients before first prosthesis surgery
Other: Autopsy — Dead patients will be autopsied: hair, urine, blood, peri-prosthetic tissue and viscera (liver, kidney, spleen, brain, heart, lung) sampling for each autopsy.
  Arms: Dead patients IMD holders autopsied; Dead patients non-IMD holders autopsied

SUMMARY:
The main objective of this study is to evaluate the systemic impact of salting out of trace elements (TE) by metallic and nonmetallic implantable medical devices (IMD) and in particular the immune response of the organism to these trace elements and of their target organs, and to identify circulating protein biomarkers which might indicate an evolution of inflammation caused by an IMD.

DETAILED DESCRIPTION:
As secondary objectives, the study aims:

* to establish the norms of concentrations of free TE and nanoparticles for some forty of elements (in particular Chrome, Cobalt, Nickel, Titanium, Tantalum, Zirconium, Tungsten, Gold, Silver, Mercury, Molybdenum, Strontium ...) in different materials (blood, urine, hair and the viscera), with non-IMD holder subjects, before and after mineralization of these materials (dead patients and autopsied non-IMD holder subjects and subjects before placement of IMD.
* to evaluate the distribution of concentrations of metals in the same materials and in peri-prothetic environment with IMD holder subjects (dead autopsied patients), more often with no inflammatory sign, with possibility of some probably inflammatory IMD.
* to evaluate the parameters of distributions of concentrations of metals in same materials (with the exception of the viscera) with living IMD holder patients, with inflammatory reaction (during revision surgery).
* to define the most suitable material (accessibility, concentrations, absence of contamination) for follow-up and evolution of inflammation in order to determinate norms of studied metals concentration.
* to determinate proportion between different forms of circulation: particulate form (analysis after full mineralization) or free form (analysis without mineralization, permitting measurement of free forms), trace elements in organism.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient subjects for re-intervention of: hip prosthesis made by ceramic-on-ceramic or metal-on-metal, hip prosthesis made by stainless steel ball and knee prosthesis made by polyethylene-on-metal;
* Autopsied patients with and without IMD;
* Covered by a health insurance.

Exclusion Criteria:

* Infection caused by prosthesis resumption;
* Professional exposure to metals;
* Patient under guardianship.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Immunophenotyping of inflammatory cells activated in contact with trace element nanoparticles | through study completion, an average of 2 years
  Demonstration of systemic inflammation induced by the trace elements existing in IMD with blood and tissue criteria:
  1/ A measure by flow cytometry to identify hyperactivated circulating mononuclear cells (macrophages, dendritic cells, T and B lymphocytes), in contact with trace element nanoparticles and thus, to highlight an immunophenotype of this inflammation.
Identification of specific circulating proteins (biomarkers) of inflammation related to trace element release | through study completion, an average of 2 years
  Demonstration of systemic inflammation induced by the trace elements existing in IMD with blood and tissue criteria:
  2/ A measure by multiplex LuminexTM (Bio-plex ProTM human inflammation panel, Bio-rad) to identify specific circulating proteins such as TNF, IFN, cytokines, chemokines, metalloproteins, related to activation of the cells of inflammation throughout release of particles and salting out of trace elements by IMD
Macroscopic characterization of tissue inflammation of autopsied patients | through study completion, an average of 2 years
  Demonstration of systemic inflammation induced by the trace elements existing in IMD with blood and tissue criteria:
  - 3/ A macroscopic study of organs to determine the possible presence of tumor foci
Microscopic characterization of tissue inflammation of autopsied patients | through study completion, an average of 2 years
  Demonstration of systemic inflammation induced by the trace elements existing in IMD with blood and tissue criteria:
  - 4/ Cytopathological analysis on slides, after sampling, fixation, inclusion and staining with hematoxylin-eosin-saffron to evaluate semi-quantitatively the type of inflammation (chronic if mononuclear cells or acute if neutrophils) and degree according to the number of inflammatory cells

SECONDARY OUTCOMES:
Trace elements dosing in liquids and tissues | through study completion, an average of 2 years
  Trace elements dosing in liquids and tissue by high resolution ICP mass spectrometry in studied sub-population (autopsied IMD holder and non-holder dead subjects, IMD holder living patients with inflammatory reaction and will undergo re-intervention) and in each analyzed material in non-mineralized form, in order to determinate concentrations of free trace elements and after full mineralization to determinate the concentrations of trace elements in nanoparticle form.
Comparison of concentrations of 40 analyzed trace elements | through study completion, an average of 2 years
  Comparison of concentrations of 40 analyzed trace elements in different materials, depending on the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Alvarez, MD, PhD, Principal Investigator — Laboratoire de Pharmacologie-Toxicologie, Hôpital Raymond Poincaré, Garches; Thomas BAUER, MD, PhD, Study Director — Orthopédie et traumatologie, Hôpital Ambroise Paré, Boulogne-Billancourt
Locations (1):
- Service de Chirurgie orthopédique, Hôpital Raymond Poincaré, Garches, Hauts-des-Seine, France

IPD SHARING:
Plan to Share IPD: No